CLINICAL TRIAL: NCT00326521
Title: Evaluation of Intrapartum Fever in Patients Receiving Epidural Anesthesia
Brief Title: Evaluation of Fever Occurring in Labor in Patients Receiving Epidural Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MemorialCare (Other)
Responsible Party: Christine Preslicka, Department of Obstetrics and Gynecology, Division of Maternal Fetal Medicine
Other Study IDs: 297-05
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Fever
Keywords: Pregnant Women; Epidural Anesthesia; Fever; Chorioamnionitis; Intrauterine pressure catheter; Pregnancy
MeSH Terms: conditions — Fever; Chorioamnionitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal serum, amniotic fluid, and umbilical cord blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Briefly, the investigators propose to evaluate nulliparous (first time mothers) patients beyond 36 0/7 weeks' gestation in active labor who already have received epidural anesthesia and have an intrauterine pressure catheter (IUPC) in place. Any patient who then develops a single temperature elevation of > 38 degrees will be eligible for inclusion and consented for the study. Maternal blood will be drawn immediately, one hour later and at delivery. Amniotic fluid will be aspirated from the pressure catheter; the first 1-2 cc will be discarded and the remainder will be evaluated for gram stain, culture, glucose level, interleukin-6 (IL-6), and proteomics. All placentas will be sent for routine pathologic examination. Cord blood will be obtained at birth for routine studies. Both maternal and cord blood will be sent for proteomic evaluation (defined). The patients with amniotic fluid that has a positive gram stain and culture will be defined as the infected group, and the patients with amniotic fluid that has a negative gram stain and culture will be defined as the uninfected group. Differences in clinical presentation and laboratory assessments, including proteomics, will be compared between the two groups to determine if there are any markers that might prove to be useful in distinguishing between these two entities (epidural fever with and without actual infection).

DETAILED DESCRIPTION:
Historically the diagnosis of chorioamnionitis (an infection of the membranes surrounding the fetus) for patients in labor has been made on the basis of multiple clinical variables such as maternal fever, fetal tachycardia, uterine tenderness, or foul smelling vaginal discharge. The diagnosis also takes into account a clinical picture consistent with risk factors such as prolonged labor and prolonged rupture of membranes. Since most of these findings are not specific, chorioamnionitis becomes the diagnosis of exclusion unless there is another explanation for the fever. Randomized studies have clearly shown that maternal antibiotics and neonatal septic work-ups are indicated once the diagnosis of chorioamnionitis has been made. Neonatal sepsis is a severe infection of the blood stream. Such policies have important implications for health care providers, on the impact of medical costs, and on the duration of hospital stay. This becomes especially true for the newborn that is transferred to the neonatal intensive care unit (NICU) for sepsis evaluation. Often times, these newborns are prophylactically treated with antibiotics based on the suspicion of an infection, while waiting for finalized blood culture results. Since newborn sepsis is such a difficult diagnosis to make, many more newborns are treated than actually have the disease and the length of their hospital stay may be significantly increased.

Over the past 15 years, both observational and randomized trials have observed an increase in maternal fever associated with epidural anesthesia in labor. These trials have shown increased ranges from 10 - 15% over baseline rates and an increased relative risk of 1.5 to 15 fold, and even up to 70 fold in one study, over the rates seen in women not receiving epidural anesthesia. After correcting for duration of labor and other confounding variables, these increases remained present. Since epidural fever is virtually impossible to distinguish from chorioamnionitis-related fever, these women are almost all treated with antibiotics and given the diagnosis of infection. This approach also has tremendous impact on the evaluation and care of the newborn. Two specific studies evaluated this impact on the neonate. Lieberman found that babies of mothers given epidural anesthesia were more likely to be evaluated for sepsis (34 vs. 9%) and treated with antibiotics (15 vs. 4%). Similarly, Philips found the same increase (25 vs. 16% and 19 vs. 11%). Both studies had very low rates of confirmed neonatal sepsis. On a national basis, the cost of this confusion nationally is tremendous.

There is one known way to distinguish between true chorioamnionitis in labor and non-infectious fever due to the epidural anesthesia. Gibbs and colleagues found that amniotic fluid aspirated from an intrauterine pressure catheter, a device commonly utilized for monitoring contractions in labor, could be used to accurately make the diagnosis of infection using gram stain and culture. More recently, many papers have shown that low glucose levels and elevated IL-6 in amniotic fluid were also accurate tests for infection. While these markers could in theory be used for distinguishing between epidural fever and true chorioamnionitis, most patients do not require such a device and this approach would not likely gain widespread favor. Alternatively, however, this approach could be used as a research tool in women who already have such a catheter in place to determine if there are additional non-invasive clinical or laboratory markers to distinguish one from the other.

Recently proteomic assessment has become an extremely effective tool in determining if there are certain markers for various diseases. Proteomics is the determination of the structure, function, and expression of all of the corresponding proteins that are encoded within the genome structure. It can also be defined as the "fingerprint" of a disease process. It involves running tandem mass spectometry on the fluid of interest. Such an approach could be extremely valuable both in determining whether the mother actually has chorioamnionitis and, if so, whether there are better markers for neonatal sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Maternal age > 18 years of age
* Estimated gestational age (EGA) > 36 0/7 weeks
* Active labor (> 4 cm dilated)
* Epidural anesthesia
* IUPC in place prior to development of fever
* Temperature of > 38 degrees
* Consents to study

Exclusion Criteria:

* Multiparous
* Maternal age < 18 years of age
* External tocometer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women >18 years of age that present to labor and delivery and are in active labor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Study Completion 2009-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Nageotte, MD, Principal Investigator — Memorial Care
Locations (2):
- United States (2):
  - Long Beach Memorial Medical Center, Long Beach, California
  - UCI Medical Center, Orange, California

REFERENCES:
- [Background] Gibbs RS, Blanco JD, St Clair PJ, Castaneda YS. Quantitative bacteriology of amniotic fluid from women with clinical intraamniotic infection at term. J Infect Dis. 1982 Jan;145(1):1-8. doi: 10.1093/infdis/145.1.1. PMID 7033397
- [Background] Lieberman E, O'donoghue C. Unintended effects of epidural analgesia during labor: a systematic review. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S31-68. doi: 10.1067/mob.2002.122522. PMID 12011872
- [Background] Ramin SM, Gambling DR, Lucas MJ, Sharma SK, Sidawi JE, Leveno KJ. Randomized trial of epidural versus intravenous analgesia during labor. Obstet Gynecol. 1995 Nov;86(5):783-9. doi: 10.1016/0029-7844(95)00269-w. PMID 7566849
- [Background] Yancey MK, Zhang J, Schwarz J, Dietrich CS 3rd, Klebanoff M. Labor epidural analgesia and intrapartum maternal hyperthermia. Obstet Gynecol. 2001 Nov;98(5 Pt 1):763-70. doi: 10.1016/s0029-7844(01)01537-x. PMID 11704166
- [Background] Lieberman E, Lang JM, Frigoletto F Jr, Richardson DK, Ringer SA, Cohen A. Epidural analgesia, intrapartum fever, and neonatal sepsis evaluation. Pediatrics. 1997 Mar;99(3):415-9. doi: 10.1542/peds.99.3.415. PMID 9041298
- [Background] Chen KT, Ringer S, Cohen AP, Lieberman E. The role of intrapartum fever in identifying asymptomatic term neonates with early-onset neonatal sepsis. J Perinatol. 2002 Dec;22(8):653-7. doi: 10.1038/sj.jp.7210818. PMID 12478449